CLINICAL TRIAL: NCT04051268
Title: Immunogenicity and Safety of Vi-DT Typhoid Conjugate Vaccine (Bio Farma) in Adults, Children and Infants, Lot to Lot Consistency, Non-inferiority to PQed (Prequalified) TCV (Typhoid Conjugate Vaccine)
Brief Title: Immunogenicity and Safety of Vi-DT (Diphtheria Toxoid) Typhoid Conjugate Vaccine (Phase III)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Typhoid 0319
Record Dates: First submitted 2019-08-06; First posted 2019-08-09 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Safety Issues; Immunogenicity
Keywords: Vaccine; Typhoid Conjugate Vaccine
MeSH Terms: interventions — Vi polysaccharide vaccine, typhoid

STUDY DESIGN:
Intervention Model Description: Subjects 6 months - 45 years of age: Randomized, observer blind, lot to lot consistency, non inferiority to PQed typhoid conjugate vaccine Subjects 46 - 60 years of age: Randomized, observer blind, lot to lot consistency, superiority to Vi polysaccharide vaccine.
  Subjects 6 months - 60 years old: Randomized, observer blind, lot to lot consistency
Who Masked: Participant, Investigator
Masking Description: Investigational Product and Active Comparator was masking Number of lot was masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Vi-DT TCV Batch 1 (Experimental): 1 dose of 0.5 ml of Vi-DT TCV vaccine batch 1
  Interventions: Biological: Vi-DT Typhoid Conjugate Vaccine
- Vi-DT TCV Batch 2 (Experimental): 1 dose of 0.5 ml of Vi-DT TCV vaccine batch 2
  Interventions: Biological: Vi-DT Typhoid Conjugate Vaccine
- Vi-DT TCV Batch 3 (Experimental): 1 dose of 0.5 ml of Vi-DT TCV vaccine batch 3
  Interventions: Biological: Vi-DT Typhoid Conjugate Vaccine
- PQed Typhoid Conjugate Vaccine (subjects 6 mo-45 yo) (Active Comparator): 1 dose of 0.5 ml of PQed TCV Vaccine
  Interventions: Biological: PQed Typhoid Conjugate Vaccine
- Vi Polysaccharide Vaccine (subjects 46-60 years old) (Active Comparator): 1 dose of 0.5 ml of Vi Polysaccharide Vaccine
  Interventions: Biological: Vi Polysaccharide Vaccine

INTERVENTIONS:
Biological: Vi-DT Typhoid Conjugate Vaccine — 1 dose of Investigational Product
  Arms: Vi-DT TCV Batch 1; Vi-DT TCV Batch 2; Vi-DT TCV Batch 3
Biological: PQed Typhoid Conjugate Vaccine — 1 dose of Active Comparator
  Arms: PQed Typhoid Conjugate Vaccine (subjects 6 mo-45 yo)
Biological: Vi Polysaccharide Vaccine — 1 dose of Active Comparator
  Arms: Vi Polysaccharide Vaccine (subjects 46-60 years old)

SUMMARY:
Phase III study, Randomized, observer blind, lot to lot consistency, non inferiority to PQed typhoid conjugate vaccine and Typhoid Vi polysaccharide vaccine.

DETAILED DESCRIPTION:
Phase III study, Randomized, observer blind, lot to lot consistency, non inferiority to PQed typhoid conjugate vaccine and to Typhoid Vi polysaccharide vaccine.

Involved participants aged 6 months old to 60 years old.

ELIGIBILITY:
Inclusion Criteria:

* Healthy.
* Subject/Parents/legal guardian(s) have been informed properly regarding the study and signed the informed consent form/and informed assent form.
* Subject/parents/legal guardian(s) will commit to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

* Subject concomitantly enrolled or scheduled to be enrolled in another trial.
* Evolving mild, moderate or severe illness, especially infectious diseases or fever (axilary temperature ³ 37.5°C).
* Known history of allergy to any component of the vaccines.
* History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection.
* Subject who has received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products, corticosteroid therapy and other immunosuppressants)
* Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives.
* Pregnancy & lactation (Adults).
* Individuals who have previously received any vaccines against typhoid fever.
* Subjects already vaccinated with any vaccine within one month prior and expect to receive other vaccines within one month following vaccination except MR (Measles Rubella) vaccine.
* Individuals who have a previously ascertained typhoid fever by laboratory confirmation (blood culture/new rapid test) at any time.
* Subject planning to move from the study area before the end of study period.

Ages: 6 Months to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3071 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | 28 days
  Seroconversion following vaccination with one dose of Vi-DT (Bio Farma) in adults, children and infants.

SECONDARY OUTCOMES:
Describe antibody response following vaccination | 28 days
  Comparison of GMT, seroconversion between each lot number of Vi-DT (Bio Farma ) vaccine in each group.
Adverse event, solicited or unsolicited | 28 days
  Number and percentage with at least one adverse event, solicited or unsolicited, within 30 minutes, 72 hours, 7 days, and 28 days after vaccination.
Comparison the safety and immunogenicity | 28 days
  Comparison of adverse events occuring until 28 days after vaccination between each lot number of Vi-DT (Bio Farma ) vaccine and PQed typhoid conjugate vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Bernie E Medise, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Jatinegara Primary Health Care, Jakarta, Jakart, Indonesia

IPD SHARING:
Plan to Share IPD: No